CLINICAL TRIAL: NCT01002846
Title: Effects of Acupuncture at ST36 and PC6 on Blood Pressure and Endothelial
Brief Title: Effects of Acupuncture at ST36 and PC6 on Blood Pressure and Endothelial Dysfunction in Hypertensive Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Oriental Medicine of Stroke & Neurological Disorders Center, Oriental Medicine of Stroke & Neurological Disorders Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMC/5H/IRB/2009/007
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Hypertension
Keywords: Efficacy; Acupuncture; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional acupuncture (Experimental): Procedure : ST 36 and PC 6 are selected, subject will undergo 20minute sessions twice a week for 8weeks. Disposable acupuncture needle(4cm sterilized stainless steel) will be inserted up to 1 cm depth
  Interventions: Procedure: acupuncture
- sham acupuncture (Sham Comparator): Procedure : Beside 1cm of ST 36 and PC 6 are selected( not meridian point), subject will undergo 20 minute. Disposable acupuncture needle(4cm sterilized stainless steel) will be inserted under 1 cm slightly.
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — acupuncture group : subject will undergo 20minute sessions twice a week for 8weeks. Disposable acupuncture needle(4cm sterilized stainless steel) will be inserted up to 1 cm depth sham acupuncture group : subject will undergo 20 minute. Disposable acupuncture needle(4cm sterilized stainless steel) will be inserted under 1 cm slightly.

SUMMARY:
This is randomised, controlled study about effects of acupuncture on blood pressure and endothelial dysfunction in stage I hypertension patient without medication. Subject will receive 8 weeks of either acupuncture or sham acupuncture, measuring FMD and blood test before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-70 diagnosed stage I hypertension ( JNC-7) without taking hypertensive medication

Exclusion Criteria:

* Secondary hypertension
* DM
* History of cardiovascular disease
* Taking hypertensive medication
* Taking hyperlipidemic medication
* Smoking
* Pregnancy or feeding woman
* Cannot follow indication or there is no agreement of patient and conservator
* Investigator decide Inappropriate to trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
To assess effects of acupuncture on endothelial function with FMD variation after 8 weeks treatments. | 8 weeks

SECONDARY OUTCOMES:
To examine the effects of acupuncture on blood pressure, lipid , hsCRP level variation with ABPM after 8 weeks treatments. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SeongUk Park, OMD, Principal Investigator — Oriental medicine center of Stroke and Neurology
Locations (1):
- Oriental Medicine of Stroke and Nerologic center, Seoul, South Korea, South Korea